CLINICAL TRIAL: NCT04991298
Title: Efficacy of the Intravenous Formulation of Fentanyl Citrate Administered Orally as Premedication in Paediatric Patients Undergoing Open Cardiac Surgery
Brief Title: Efficacy of iv Fentanyl Citrate Administered Oral as a Pediatric Premedication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ibrahim Mabrouk Ibrahim, Assistant lecturer, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124
Record Dates: First submitted 2021-05-27; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Premedication; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): patients will be premedicated with the undiluted IV formulation of Midazolam
  Interventions: Drug: Oral premedication
- Group F (Active Comparator): patients will be premedicated with the undiluted IV formulation of fentanyl citrate
  Interventions: Drug: Oral premedication

INTERVENTIONS:
Drug: Oral premedication — Oral anesthesia premedication for congenital Cardiac surgery
  Other Names: Midazolam , fentanyl

SUMMARY:
evaluate the efficacy of the intravenous formulation of fentanyl citrate administered orally as a sedative premedication, we will compare it with oral midazolam, as a gold standard premedication, in paediatric congenital cardiac surgeries

DETAILED DESCRIPTION:
In this double-blinded randomized controlled study, after approval by the local ethics committee, paediatric patients, aged 1 to 7 years, scheduled for elective surgical procedures for correction of congenital heart disease will be enrolled. Patients with hepatic or renal disorders, gastrointestinal tract disorders or malformation, conduction disorders, coronary artery disease, emergency operations, mental disabilities, and known reactions to the drugs to be used will be excluded. After assessing the patient for anaesthesia, informed consent of patients about study and anaesthesia will be obtained.Children will be kept off solid food for 6 hours and of clear fluids for 2 hours. The premedication will be administered orally mixed with equal volume of 5% dextrose and using a 5-ml syringe, 30 minutes before admission to operating room by a member of the nursing staff unaware of the group allocation, in the preoperative holding area, in the presence of one parent. A randomized block design will be used for allocation of patients into two groups (50 patients each); one group of patients will receive midazolam (Group M) and the other will receive fentanyl (Group F) as a sedative premedication.

1. Group M: patients will be premedicated with the undiluted IV formulation of Midazolam (5 mg/mL), 0.5 mg/kg up to 15 mg per patient. The dose is chosen to be similar to the dose of midazolam used in other previous studies ().
2. Group F: patients will be premedicated with the undiluted IV formulation of fentanyl citrate (50 µg/mL), 10 µg/kg up to 400 µg per patient. The dose is chosen to be similar to the dose of OTFC used in other previous studies

ELIGIBILITY:
Inclusion Criteria:

* paediatric congenital heart disease patients, aged 1 to 7 years, scheduled for elective surgical procedures for correction of congenital heart disease

Exclusion Criteria:

* Patients with hepatic or renal disorders, gastrointestinal tract disorders or malformation, conduction disorders, coronary artery disease, emergency operations, mental disabilities, and known reactions to the drugs to be used will be excluded.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Patient's acceptance of the medication (score from 1 to 3) | 1 year
  Response of the child to acceptance of premedication will be assessed on a three-point scale:
  1. = Spits/vomits the premedication.
  2. = Accepts it/but dislikes the taste.
  3. = Accepts it/likes the taste.
Reaction to separation from parents (score from 1 to 4) | 1 year
  The response of the children when taken away from the parents will be recorded as the end point of premedication. It will be assessed on a four point scale:
  1. = Inconsolable cry.
  2. = Complaining.
  3. = Quiet but awake.
  4. = Sleepy.
Sedation score ( score from 1 to 6) | 1 year
  The degree of sedation, when the child will be first seen in the operating room (OR), will be scaled from 1 to 6 according to the Ramsay Sedation Scale.
  1. =Anxious and agitated or restless, or both.
  2. =Cooperative, oriented, and calm.
  3. =Responsive to commands only.
  4. =Exhibiting brisk response to light glabellar tap or loud auditory stimulus.
  5. =Exhibiting a sluggish response to light glabellar tap or loud auditory stimulus.
  6. =Unresponsive.
Ease of Induction of general anaesthesia (score from 1 to 4) | 1 year
  A 4-point scoring system will used to evaluate the child's behaviour at anaesthesia induction and mask acceptance
  1= Calm and cooperating 2 =Anxious but without resistance 3 =Anxious with slight resistance 4 =Crying and/or struggling against mask

SECONDARY OUTCOMES:
Hemodynamic effects | 1 year
  Heart rate (beats/min)
Adverse effects | 1 year
  nausea, vomiting, illusion, pruritis, paradoxical hyperactive reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No